CLINICAL TRIAL: NCT00970801
Title: Identification of Host Susceptibility Factors and Development of Biomarkers for Diagnosis, Prognosis and Treatment of Nontuberculous Mycobacterial Lung Disease
Brief Title: Study of Nontuberculous Mycobacterial Lung Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won-Jung Koh, MD, Samsung Medical Center
Other Study IDs: 2008-09-016
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Nontuberculous Mycobacterial Lung Disease
Keywords: Atypical mycobacteria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The incidence of pulmonary disease caused by nontuberculous mycobacteria (NTM) has been increasing, and a substantial proportion of these patients have no preexisting lung disease and no demonstrable immunodeficiency. These patients are predominantly nonsmoking elderly women. High-resolution computed tomography scans revealed the characteristic findings of multifocal bronchiectasis combined with multiple small nodules. NTMs are ubiquitous environmental organisms. Because exposure to these organisms is universal and the occurrence of the disease is rare, normal host defense mechanisms must be effective enough to prevent the infection.

All patients with NTM lung disease do not need to receive long-term antibiotic treatment. As the American Thoracic Society guidelines point out, one of the most difficult questions may be when to start antibiotic therapy in patients with NTM lung disease. The decision to begin treatment is made by weighing the anticipated benefits and risks. The decision is relatively easy in patients with profound symptoms and destructive lesions; however, the decision is difficult in patients with mild symptoms and non-advanced lesions. Factors that must be considered include the patients' age, whether the symptoms are mild or equivocal, and the presence of comorbidities. In all cases, close observation is necessary if treatment is not performed. However, few studies have shown that patients with certain characteristics show disease progression.

The treatment of NTM pulmonary disease depends on the infecting species, but decisions concerning the institution of treatment are never easy. Treatment requires the use of multiple drugs for 18 to 24 months. Thus, treatment is expensive, often has significant side effects, and is frequently not curative. Therefore, clinicians should be confident that there is sufficient pathology to warrant prolonged, multidrug treatment regimens. In all of the situations, outcomes can be best optimized only when clinicians, radiologists, and laboratories work cooperatively.

This study will examine why some people are more susceptible to NTM lung disease and why some people of NTM lung disease are more difficult to treat. This study will examine the patient and bacterial characteristics, course of disease and treatment of NTM infections, as well as the genetics involved in these infections.

Patients with diagnosed NTM lung disease may be eligible for this study. All participants will have a medical and family history, blood tests, imaging studies that may include X-rays, computed tomography (CT) scans, and genetic and serologic studies. The aim of this study is to identify patient and bacterial characteristics that contribute to disease susceptibility, disease progression, and treatment failure. Subjects are recruited from among patients who are diagnosed to have NTM lung disease at the Samsung Medical Center in the Republic of Korea.

ELIGIBILITY:
Inclusion Criteria:

* Patients who fulfill the diagnostic criteria of NTM lung disease

Exclusion Criteria:

* Non-applicable

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients visited Samsung Medical Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2008-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | weekly

SECONDARY OUTCOMES:
disease susceptibility, disease progression, treatment failure | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Won-Jung Koh, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim BG, Kang N, Kim SY, Kim DH, Kim H, Kwon OJ, Huh HJ, Lee NY, Jhun BW. The lung microbiota in nontuberculous mycobacterial pulmonary disease. PLoS One. 2023 May 26;18(5):e0285143. doi: 10.1371/journal.pone.0285143. eCollection 2023. PMID 37235629
- [Derived] Kang N, Jeon K, Kim H, Kwon OJ, Huh HJ, Lee NY, Daley CL, Koh WJ, Jhun BW. Outcomes of Inhaled Amikacin-Containing Multidrug Regimens for Mycobacterium abscessus Pulmonary Disease. Chest. 2021 Aug;160(2):436-445. doi: 10.1016/j.chest.2021.02.025. Epub 2021 Feb 20. PMID 33621600
- [Derived] Jhun BW, Moon SM, Jeon K, Kwon OJ, Yoo H, Carriere KC, Huh HJ, Lee NY, Shin SJ, Daley CL, Koh WJ. Prognostic factors associated with long-term mortality in 1445 patients with nontuberculous mycobacterial pulmonary disease: a 15-year follow-up study. Eur Respir J. 2020 Jan 2;55(1):1900798. doi: 10.1183/13993003.00798-2019. Print 2020 Jan. PMID 31619468
- [Derived] Jhun BW, Kim SY, Moon SM, Jeon K, Kwon OJ, Huh HJ, Ki CS, Lee NY, Shin SJ, Daley CL, Koh WJ. Development of Macrolide Resistance and Reinfection in Refractory Mycobacterium avium Complex Lung Disease. Am J Respir Crit Care Med. 2018 Nov 15;198(10):1322-1330. doi: 10.1164/rccm.201802-0321OC. PMID 29877739
- [Derived] Koh WJ, Jeong BH, Kim SY, Jeon K, Park KU, Jhun BW, Lee H, Park HY, Kim DH, Huh HJ, Ki CS, Lee NY, Kim HK, Choi YS, Kim J, Lee SH, Kim CK, Shin SJ, Daley CL, Kim H, Kwon OJ. Mycobacterial Characteristics and Treatment Outcomes in Mycobacterium abscessus Lung Disease. Clin Infect Dis. 2017 Feb 1;64(3):309-316. doi: 10.1093/cid/ciw724. Epub 2016 Nov 10. PMID 28011608
- [Derived] Jeong BH, Jeon K, Park HY, Moon SM, Kim SY, Lee SY, Shin SJ, Daley CL, Koh WJ. Peak Plasma Concentration of Azithromycin and Treatment Responses in Mycobacterium avium Complex Lung Disease. Antimicrob Agents Chemother. 2016 Sep 23;60(10):6076-83. doi: 10.1128/AAC.00770-16. Print 2016 Oct. PMID 27480854
- [Derived] Koh WJ, Jeong BH, Jeon K, Kim SY, Park KU, Park HY, Huh HJ, Ki CS, Lee NY, Lee SH, Kim CK, Daley CL, Shin SJ, Kim H, Kwon OJ. Oral Macrolide Therapy Following Short-term Combination Antibiotic Treatment of Mycobacterium massiliense Lung Disease. Chest. 2016 Dec;150(6):1211-1221. doi: 10.1016/j.chest.2016.05.003. Epub 2016 May 7. PMID 27167209
- [Derived] Jeong BH, Jeon K, Park HY, Kim SY, Lee KS, Huh HJ, Ki CS, Lee NY, Shin SJ, Daley CL, Koh WJ. Intermittent antibiotic therapy for nodular bronchiectatic Mycobacterium avium complex lung disease. Am J Respir Crit Care Med. 2015 Jan 1;191(1):96-103. doi: 10.1164/rccm.201408-1545OC. PMID 25393520
- [Derived] Jeong BH, Kim SY, Jeon K, Lee SY, Shin SJ, Koh WJ. Serodiagnosis of Mycobacterium avium complex and Mycobacterium abscessus complex pulmonary disease by use of IgA antibodies to glycopeptidolipid core antigen. J Clin Microbiol. 2013 Aug;51(8):2747-9. doi: 10.1128/JCM.00702-13. Epub 2013 Jun 5. PMID 23740728
- [Derived] Kim SY, Lee ST, Jeong BH, Park HY, Jeon K, Kim JW, Shin SJ, Koh WJ. Genotyping of Mycobacterium intracellulare isolates and clinical characteristics of lung disease. Int J Tuberc Lung Dis. 2013 May;17(5):669-75. doi: 10.5588/ijtld.12.0575. PMID 23575334